CLINICAL TRIAL: NCT02448810
Title: A Phase 2a Randomized, Open-label Study to Assess the Safety, Tolerability, and Efficacy of BAX69 in Combination With 5-FU/Leucovorin or Panitumumab Versus Standard of Care in Subjects With Metastatic Colorectal Cancer
Brief Title: Phase 2a Study of BAX69 and 5-FU/Leucovorin or Panitumumab Versus Standard of Care in Subjects With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on overall benefit-risk assessment.
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 391401; 2015-000896-28 (EudraCT Number)
Record Dates: First submitted 2015-05-15; First posted 2015-05-20 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Part 1: Subjects with mutated tumor (mt) (KRAS or NRAS) (Experimental): Subjects stratified according to their mutation status.
  Interventions: Biological: BAX69 + infusional 5-FU/LV
- Part 1: Subjects with wild-type (wt) tumor (KRAS and NRAS wt) (Experimental): Subjects stratified according to their mutation status.
  Interventions: Biological: BAX69 + panitumumab
- Part 2: Subjects with KRAS or NRAS mutated (Experimental): Subjects stratified according to their mutation status.
  Interventions: Biological: BAX69 + 5-FU/LV
- Part 2: Subjects with KRAS and NRAS wt tumor (Experimental): Subjects stratified according to their mutation status.
  Interventions: Biological: BAX69 + panitumumab
- Part 2: Standard of Care- Subjects with KRAS or NRAS mutated (Active Comparator): Subjects stratified according to their mutation status.
  Interventions: Drug: Standard of Care
- Part 2: Standard of Care- Subjects with KRAS and NRAS wt tumor (Active Comparator): Subjects stratified according to their mutation status.Subjects stratified according to their mutation status.
  Interventions: Biological: Standard of Care

INTERVENTIONS:
Biological: BAX69 + infusional 5-FU/LV — Study Part 1: Safety Run-in
  * Administered weekly as part of a 4 week treatment cycle
  * Intravenous injection
  Other Names: Macrophage Migration Inhibitory Factor Antibody (Anti-MIF); Imalumab
  Arms: Part 1: Subjects with mutated tumor (mt) (KRAS or NRAS)
Biological: BAX69 + panitumumab — Study Part 1: Safety Run-in
  * Administered weekly as part of a 4 week treatment cycle
  * Intravenous injection
  Other Names: Imalumab; Anti-MIF
  Arms: Part 1: Subjects with wild-type (wt) tumor (KRAS and NRAS wt)
Biological: BAX69 + 5-FU/LV — Study Part 2: Administered weekly as part of a 4 week treatment cycle
  •Intravenous injection
  Other Names: Imalumab; Anti-MIF
  Arms: Part 2: Subjects with KRAS or NRAS mutated
Biological: BAX69 + panitumumab — Study Part 2: Administered weekly as part of a 4 week treatment cycle
  •Intravenous injection
  Other Names: Imalumab; Anti-MIF
  Arms: Part 2: Subjects with KRAS and NRAS wt tumor
Drug: Standard of Care — * Investigator's choice
  * Dose according to drug label
  Arms: Part 2: Standard of Care- Subjects with KRAS or NRAS mutated
Biological: Standard of Care — * Investigator's choice
  * Dose according to drug label
  * Choice includes panitumumab in KRAS &NRAS wt group only
  Arms: Part 2: Standard of Care- Subjects with KRAS and NRAS wt tumor

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of BAX69 in combination with 5-fluorouracil (5-FU)/leucovorin (LV) or panitumumab to determine the recommended phase II dose (RP2D) of each combination; and to compare the efficacy between BAX69 in combination with 5-FU/LV for subjects with KRAS or NRAS mutated tumor (mt) or panitumumab, for subjects with KRAS and NRAS wild type tumor (wt) and standard of care (SoC) per investigator choice as third or fourth treatment line in subjects with progressive measurable metastatic colorectal cancer (mCRC).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a signed informed consent
2. Male and female subjects 18 years of age and older at the time of screening
3. Subjects who progressed after receiving at least 2, but no more than 3, prior SoC treatment lines
4. Anticipated life expectancy >3 months at the time of screening
5. Weight between 40 kg and 180 kg
6. Histologically or cytologically confirmed diagnosis of CRC
7. Metastatic CRC not amenable to surgical resection
8. Known KRAS and NRAS mutation status (if unknown status for either of these genes, and no archival tissues is available, a fresh tumor biopsy will be made)
9. At least 1 measurable lesion as defined by RECIST v1.1
10. ECOG PS of 0-2
11. Adequate hematological function, defined as:

    1. Platelet count ≥ 100,000/μL
    2. Prothrombin time and activated partial thromboplastin time (aPTT) < 1.5 times the upper limit of normal (ULN)
    3. Absolute neutrophil count (ANC) ≥ 1,000/μL
    4. Hemoglobin ≥ 9 g/dL, without the need for transfusion in the 2 weeks prior to screening
12. Adequate renal function, defined as serum creatinine ≤ 2.0 times ULN and creatinine clearance > 50 mL/min
13. Adequate liver function, defined as:

    1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)

       ≤ 2.5 times ULN for subjects without liver metastases, or ≤ 5 times ULN in the presence of liver metastases
    2. Bilirubin ≤ 2.0 times ULN, unless subject has known Gilbert's syndrome
14. Adequate venous access
15. For female subjects of childbearing potential, the subject presents with a negative serum pregnancy test at screening and agrees to employ 2 forms of adequate birth control measures, including at least 1 barrier method (eg, diaphragm with spermicidal jelly or foam, or [for male partner] condom) throughout the course of the study and for at least 90 days after the last administration of BAX69. Other acceptable contraceptive measures include birth control pills/patches or intrauterine devices
16. For male subjects, the subject must agree to use adequate contraceptive measures including at least 1 barrier method (eg, condom with spermicidal jelly or foam and [for the female partner] diaphragm with spermicidal jelly or foam, birth control pills/patches, or intrauterine device) and abstain from sperm donation throughout the course of the study and for at least 90 days after the last administration of BAX69
17. Subject is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Known central nervous system metastases
2. Prior malignancy(s) within the past 3 years, with the exception of curatively treated basal or squamous cell carcinoma of the skin, locally advanced prostate cancer, ductal carcinoma in situ of breast, in situ cervical carcinoma and superficial bladder cancer
3. Prior treatment with panitumumab for subjects with KRAS and NRAS wt tumor
4. Residual AE from previous treatment > Grade 1
5. Prior intolerance to fluoropyrimidine for subjects with KRAS or NRAS mut tumor
6. Myocardial infarction within 6 months prior to C1D1, and/or prior diagnoses of congestive heart failure (New York Heart Association Class III or IV), unstable angina, unstable cardiac arrhythmia requiring medication; and/or the subject is at risk for polymorphic ventricular tachycardia (eg, hypokalemia, family history or long QT syndrome)
7. Uncontrolled hypertension defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg confirmed upon repeated measures
8. LVEF < 40% as determined by echocardiogram performed at screening or within 90 days prior to C1D1
9. QT/QTc interval > 450 msec, as determined by screening ECG performed no earlier than 1 week before C1D1
10. Prior anti-tumor therapy (chemotherapy, radiotherapy, antibody therapy, molecular targeted therapy, retinoid therapy or hormonal therapy) within 4 weeks prior to C1D1.
11. Major surgery within 4 weeks prior to C1D1
12. Active joint inflammation or history of inflammatory arthritis or other immune disorder involving joints
13. Active infection involving IV antibiotics within 2 weeks prior to C1D1
14. Known history of, or active hepatitis B virus (HBV), hepatitis C virus (HCV) or active tuberculosis
15. Known history of human immunodeficiency virus (HIV) type 1/2 or other immunodeficiency disease
16. Subject has received a live vaccine within 4 weeks prior to C1D1
17. Known hypersensitivity to any component of recombinant protein production by CHO cells
18. Exposure to an investigational product or investigational device in another clinical study within 4 weeks prior to C1D1, or is scheduled to participate in another clinical study involving an investigational product or device during the course of this study
19. Subject is nursing or intends to begin nursing during the course of the study
20. Any disorder or disease, or clinically significant abnormality on laboratory or other clinical test(s) (eg, blood tests, ECG), that in medical judgment of the investigator may impede the subject's participation in the study, pose increased risk to the subject, and/or confound the results of the study
21. Subject is a family member or employee of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- United States (12):
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Indiana University Health, Goshen, Indiana
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Beth Israel, New York, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - The Jones Clinic, PC, Germantown, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - CTRC at University of Texas Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 centers in the United States, the United Kingdom and Spain between 15 June 2015 (first participant first visit) and 15 February 2017 (last participant last visit).
Pre-assignment Details: Overall (part 1 and 2) 115 participants were screened, 85 participants were randomized and 79 participants were treated. In part 1, 17 participants were screened, 5 failed screening, 12 were randomized and treated. In part 2, 98 participants were screened, 17 failed screening and 8 did not start the study, 73 were randomized and 67 were treated.
Groups:
- Part 1: Imalumab 7.5 mg/kg + 5-FU/LV: Participants with mutated tumors (mutated kirsten rat sarcoma viral oncogene homolog, mutated neuroblastoma rat sarcoma viral oncogene homolog [KRAS mut, NRAS mut]) received 7.5 milligram per kilogram (mg/kg) dose of imalumab every week (QW) in combination with 5-fluorouracil/leucovorin ([FU/LV] LV 400 milligram per square meter [mg/m^2] intravenous (IV) infusion over 2 hours, followed by 5 FU 2400 mg/m^2 IV infusion over 46 hours) for every 2 weeks (Q2W) IV infusion as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
- Part 1: Imalumab 7.5 mg/kg + Panitumumab: Participants with wild-type tumors (wild type Kirsten rat sarcoma viral oncogene homolog, wild neuroblastoma rat sarcoma viral oncogene homolog [KRAS wt, NRAS wt]) received 7.5 mg/kg dose of imalumab QW in combination with panitumumab 6 mg/kg Q2W IV infusion as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
- Part 1: Imalumab 10 mg/kg + 5-FU/LV: Participants with mutated tumors (KRAS mut, NRAS mut) received 10 mg/kg dose of imalumab QW in combination with 5-FU/LV (LV 400 mg/m^2 IV infusion over 2 hours, followed by 5 FU 2400 mg/m^2 IV infusion over 46 hours) Q2W IV infusion as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
- Part 1: Imalumab 10 mg/kg + Panitumumab: Participants with wild-type tumors (KRAS wt, NRAS wt) received 10 mg/kg dose of imalumab QW in combination with panitumumab 6 mg/kg Q2W IV infusion as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
- Part 2: Imalumab 10 mg/kg + 5-FU/LV: Participants with mutated tumors (KRAS mut, NRAS mut) received 10 mg/kg dose of imalumab as a recommended phase 2 dose (RP2D) QW in combination with 5-FU/LV (LV 400 mg/m^2 IV infusion over 2 hours, followed by 5 FU 2400 mg/m^2 IV infusion over 46 hours) Q2W IV infusion as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
- Part 2: Standard of Care Mutant: Participants with mutated tumors (KRAS mut, NRAS mut) received standard of care (SoC) as chosen by the investigator and was administered in accordance to product label as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
- Part 2: Imalumab 10 mg/kg + Panitumumab: Participants with wild-type tumors (KRAS wt, NRAS wt) received 10 mg/kg dose of imalumab as a RP2D QW in combination with panitumumab 6 mg/kg Q2W IV infusion as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
- Part 2: Standard of Care Wild Type: Participants with wild-type tumors (KRAS wt, NRAS wt) received SoC as chosen by the investigator and was administered in accordance to product label as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
Period: Overall Study
Arm/Group | Part 1: Imalumab 7.5 mg/kg + 5-FU/LV | Part 1: Imalumab 7.5 mg/kg + Panitumumab | Part 1: Imalumab 10 mg/kg + 5-FU/LV | Part 1: Imalumab 10 mg/kg + Panitumumab | Part 2: Imalumab 10 mg/kg + 5-FU/LV | Part 2: Standard of Care Mutant | Part 2: Imalumab 10 mg/kg + Panitumumab | Part 2: Standard of Care Wild Type
Started | 3 | 3 | 3 | 3 | 31 | 16 | 18 | 8
Treated | 3 | 3 | 3 | 3 | 29 | 13 | 18 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 31 | 16 | 18 | 8
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 3 | 5 | 0 | 2
Not completed — Other (study terminated by sponsor) | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 1
Not completed — Death | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Other (Progressive disease) | 2 | 2 | 0 | 3 | 23 | 9 | 14 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other (unspecified) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who received at least 1 administration of study drug. Baseline was calculated only for the treated participants and not for the enrolled participants.
Groups:
- Part 1: Imalumab 7.5 mg/kg + 5-FU/LV: Participants with mutated tumors (KRAS mut, NRAS mut) received 7.5 mg/kg dose of imalumab QW in combination with 5- FU/LV (LV 400 mg/m^2 IV infusion over 2 hours, followed by 5 FU 2400 mg/m^2 IV infusion over 46 hours) for Q2W IV infusion as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
- Part 1: Imalumab 7.5 mg/kg + Panitumumab: Participants with wild-type tumors (KRAS wt, NRAS wt) received 7.5 mg/kg dose of imalumab QW in combination with panitumumab 6 mg/kg Q2W IV infusion as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Part 1: Imalumab 7.5 mg/kg + 5-FU/LV | Part 1: Imalumab 7.5 mg/kg + Panitumumab | Part 1: Imalumab 10 mg/kg + 5-FU/LV | Part 1: Imalumab 10 mg/kg + Panitumumab | Part 2: Imalumab 10 mg/kg + 5-FU/LV | Part 2: Standard of Care Mutant | Part 2: Imalumab 10 mg/kg + Panitumumab | Part 2: Standard of Care Wild Type | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 31 | 16 | 18 | 8 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 3 | 2 | 21 | 12 | 13 | 5 | 57
  >=65 years | 2 | 3 | 0 | 1 | 10 | 4 | 5 | 3 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 13 | 5 | 7 | 6 | 33
  Male | 2 | 3 | 3 | 2 | 18 | 11 | 11 | 2 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 5 | 2 | 3 | 0 | 12
  Not Hispanic or Latino | 3 | 2 | 3 | 2 | 26 | 14 | 15 | 8 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 7
  White | 2 | 3 | 3 | 2 | 26 | 14 | 18 | 6 | 74
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Progression-Free Survival (PFS)
Description: PFS was defined as time between treatment initiation and tumor progression (per Response Evaluation Criteria in Solid Tumors [RECIST] v1.1 criteria) or death from any cause, with censoring of participants who were lost to follow-up or withdrew consent.
Time Frame: From start of the study up to safety follow-up visit occurred (30 [-/+7]) days after the last dose of study treatment or until disease progression
Population: Full analysis set (FAS) included all participants who received at least 1 administration of study drug, and who had 1 postbaseline tumor response assessment based on RECIST v1.1, or died within 18 weeks of the start of treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 2: Imalumab 10 mg/kg + 5-FU/LV | Part 2: Standard of Care Mutant | Part 2: Imalumab 10 mg/kg + Panitumumab | Part 2: Standard of Care Wild Type
Number analyzed (Participants) | 29 | 12 | 18 | 7
weeks | 11.1 [8.4 to 16.1] | 8.3 [7.4 to 23.3] | 9.3 [8.1 to 24.9] | 7.3 [3.7 to NA] — Upper limit was not available.
Statistical Analysis 1: Comparison: Part 2: Imalumab 10 mg/kg + 5-FU/LV vs Part 2: Standard of Care Mutant; Test type: Other; p = 0.246, Log Rank — P-value is based on a one-sided log-rank test; Hazard Ratio (HR) = 0.8, 70% CI 2-sided [0.5 to 1.1]; Hazard Ratio and 70% CI are based on a Cox proportional hazards model with a covariate for treatment (imalumab vs SoC)
Statistical Analysis 2: Comparison: Part 2: Imalumab 10 mg/kg + Panitumumab vs Part 2: Standard of Care Wild Type; Test type: Other; p = 0.354, Log Rank — P-value is based on a one-sided log-rank test; Hazard Ratio (HR) = 0.8, 70% CI 2-sided [0.5 to 1.4]; Hazard Ratio and 70% CI are based on a Cox proportional hazards model with a covariate for treatment (imalumab vs SoC)

2. Primary Outcome: Part 1: Number of Participants With Occurrence of Dose Limiting Toxicity (DLT)
Description: DLT was defined as any drug-related treatment-emergent adverse event (TEAE) (graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v4.03) that occurs during the first 28 days after treatment start and that meets any of the following criteria: i) Any >= Grade 3 non-hematologic toxicity (excluding: mucositis/stomatitis of Grade 3; diarrhea of <3 days duration; nausea and vomiting <3 days duration; fatigue of <7 days duration; alopecia; single laboratory value out of the normal range that has no clinical significance and that resolves to <= Grade 2 with adequate measures within 7 days) ii) Any Grade 4 hematologic toxicity (excluding: grade 4 neutropenia lasting for <= 5 days; isolated grade 4 lymphocytopenia) iii) Grade 3 febrile neutropenia iv) Grade 3 thrombocytopenia associated with bleeding v) Any life-threatening complication or abnormality not covered in NCI CTCAEv4.03.
Time Frame: From start of study treatment up to 28 days
Population: SAS included all participants who received at least 1 administration of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Imalumab 7.5 mg/kg + 5-Fluorouracil/Leucovorin (FU/LV): Participants with mutated tumors (KRAS mut, NRAS mut) received 7.5 mg/kg dose of imalumab QW in combination with 5- FU/LV (LV 400 mg/m^2 IV infusion over 2 hours, followed by 5 FU 2400 mg/m^2 IV infusion over 46 hours) for Q2W IV infusion as a part of 4-week/28-day treatment cycle and continued until disease progression, unacceptable toxicity, death, or participant withdrawal of consent, whichever occurred first.
Arm/Group | Part 1: Imalumab 7.5 mg/kg + 5-Fluorouracil/Leucovorin (FU/LV) | Part 1: Imalumab 7.5 mg/kg + Panitumumab | Part 1: Imalumab 10 mg/kg + 5-FU/LV | Part 1: Imalumab 10 mg/kg + Panitumumab
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Occurrence of Binding and/or Neutralizing Anti-imalumab Antibodies
Description: Number of participants with occurrence of binding and/or neutralizing anti-imalumab antibodies were reported.
Time Frame: From start of study drug administration up to end of treatment (EOT) (approximately 21 Months)
Population: SAS included all participants who received at least 1 administration of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Imalumab 7.5 mg/kg + 5-Fluorouracil/Leucovorin (FU/LV) | Part 1: Imalumab 7.5 mg/kg + Panitumumab | Part 1: Imalumab 10 mg/kg + 5-FU/LV | Part 1: Imalumab 10 mg/kg + Panitumumab | Part 2: Imalumab 10 mg/kg + 5-FU/LV | Part 2: Standard of Care Mutant | Part 2: Imalumab 10 mg/kg + Panitumumab | Part 2: Standard of Care Wild Type
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 29 | 13 | 18 | 7
Participants
  Baseline (Binding antibody): number analyzed (Participants) | 3 | 3 | 3 | 1 | 27 | 12 | 18 | 6
  Baseline (Binding antibody) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  End of Study (Binding antibody): number analyzed (Participants) | 2 | 1 | 3 | 1 | 19 | 2 | 12 | 2
  End of Study (Binding antibody) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Baseline (Neutralizing antibody): number analyzed (Participants) | 3 | 3 | 3 | 1 | 27 | 12 | 18 | 6
  Baseline (Neutralizing antibody) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  End of Study (Neutralizing antibody): number analyzed (Participants) | 2 | 1 | 3 | 1 | 19 | 2 | 12 | 2
  End of Study (Neutralizing antibody) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Incidence of Infusion Reactions After Imalumab Administration
Description: Infusion reaction was defined as any relevant sign or symptom occurring during or after imalumab infusion and considered by the investigator as an infusion reaction.
Time Frame: From start of study drug administration up to EOT (approximately 21 Months)
Population: SAS included all participants who received at least 1 administration of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Imalumab 7.5 mg/kg + 5-Fluorouracil/Leucovorin (FU/LV) | Part 1: Imalumab 7.5 mg/kg + Panitumumab | Part 1: Imalumab 10 mg/kg + 5-FU/LV | Part 1: Imalumab 10 mg/kg + Panitumumab | Part 2: Imalumab 10 mg/kg + 5-FU/LV | Part 2: Standard of Care Mutant | Part 2: Imalumab 10 mg/kg + Panitumumab | Part 2: Standard of Care Wild Type
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 29 | 13 | 18 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any AE that results in any of the following outcomes: death, a life-threatening event, inpatient hospitalization or prolongation of an existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital anomaly/birth defect, other medically important events based upon appropriate medical judgement. TEAEs was defined as any event not present prior to the initiation of the treatments or any event already present that worsens in either intensity or frequency following exposure to the treatments.
Time Frame: From start of study drug administration up to EOT (approximately 21 Months)
Population: SAS included all participants who received at least 1 administration of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Imalumab 7.5 mg/kg + 5-Fluorouracil/Leucovorin (FU/LV) | Part 1: Imalumab 7.5 mg/kg + Panitumumab | Part 1: Imalumab 10 mg/kg + 5-FU/LV | Part 1: Imalumab 10 mg/kg + Panitumumab | Part 2: Imalumab 10 mg/kg + 5-FU/LV | Part 2: Standard of Care Mutant | Part 2: Imalumab 10 mg/kg + Panitumumab | Part 2: Standard of Care Wild Type
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 29 | 13 | 18 | 7
Participants
  SAEs | 1 | 1 | 1 | 2 | 15 | 8 | 7 | 2
  TEAEs | 3 | 3 | 3 | 3 | 28 | 13 | 17 | 7

6. Secondary Outcome: Number of Participants With Response Evaluation According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: Number of participants with response evaluation according to RECIST v1.1 was evaluated according to complete response (CR): disappearance of all target and non-target lesions and no new lesions; partial response (PR): >= 30 percent (%) decrease in the sum of diameters of target lesions (compared to baseline) and no new lesions; stable disease (SD): neither sufficient shrinkage to qualify as a response nor sufficient growth to qualify as progression; progressive disease (PD): >= 20% increase in the sum of diameters of target lesions and an absolute increase in sum of diameters of >=5 millimeter (mm) (compared to the previous minimum sum) or progression of a new lesion.
Time Frame: Day 28 of Cycle 2 followed by every 2 Cycles of 28 day Cycles: Day 56, Day 112, Day 168 and Day 224
Population: FAS included all participants who received at least 1 administration of study drug, and had 1 postbaseline tumor response assessment based on RECIST v1.1, or died within 18 weeks of the start of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Imalumab 7.5 mg/kg + 5-Fluorouracil/Leucovorin (FU/LV) | Part 1: Imalumab 7.5 mg/kg + Panitumumab | Part 1: Imalumab 10 mg/kg + 5-FU/LV | Part 1: Imalumab 10 mg/kg + Panitumumab | Part 2: Imalumab 10 mg/kg + 5-FU/LV | Part 2: Standard of Care Mutant | Part 2: Imalumab 10 mg/kg + Panitumumab | Part 2: Standard of Care Wild Type
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 29 | 12 | 18 | 7
Participants
  Best Overall Response: Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Best Overall Response: Partial Response (PR) | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1
  Best Overall Response: Stable Disease (SD) | 1 | 1 | 2 | 1 | 14 | 4 | 6 | 2
  Best Overall Response: Progressive Disease (PD) | 2 | 0 | 1 | 2 | 15 | 7 | 8 | 4
  Best Overall Response: Not Evaluable (NE) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

7. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization until death due to any cause. Here, number of participants analyzed was based on the number of participants who underwent death.
Time Frame: From start of study drug administration up to EOT (approximately 21 Months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 1: Imalumab 7.5 mg/kg + 5-Fluorouracil/Leucovorin (FU/LV) | Part 1: Imalumab 7.5 mg/kg + Panitumumab | Part 1: Imalumab 10 mg/kg + 5-FU/LV | Part 1: Imalumab 10 mg/kg + Panitumumab | Part 2: Imalumab 10 mg/kg + 5-FU/LV | Part 2: Standard of Care Mutant | Part 2: Imalumab 10 mg/kg + Panitumumab | Part 2: Standard of Care Wild Type
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 16 | 10 | 8 | 3
weeks | 24.9 [7.4 to 40.4] | 42.7 [15.4 to 77.4] | 42.7 [16.9 to 42.7] | 24.9 [9.4 to 42.1] | 31.9 [26.3 to 58.0] | 27.2 [9.3 to 46.7] | 31.4 [19.9 to NA] — The median and 95% confidence interval was not available due to insufficient number of events at the end of the study. | NA [NA to NA] — The median and 95% confidence interval was not available due to insufficient number of events at the end of the study.

8. Secondary Outcome: Change From Baseline for Quality of Life (QoL) Measure - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 was a validated instrument used to measure QoL and assess symptoms and side effects of treatment and the impact on everyday life.The QLQ-C30 was composed of: A) 5 multi-item functioning scales(physical, role, social, emotional and cognitive), that were answered on a 4-point scale (1=Not at all,2=A Little,3=Quite a Bit,4=Very Much). Each score range from 0 to 100 with a higher score representing a higher level of functioning and a better QoL. B) A global health status/QoL scale that was answered on a 7-point scale (1=Very Poor to 7=Excellent). Each score range from 0 to 100 with a higher score representing a better QoL. C) 9 symptom scales(fatigue, nausea/vomiting,pain,financial impact/difficulties,appetite loss,diarrhea, constipation,sleep disturbance/insomnia and dyspnea), that were answered on a 4-point scale (1=Not at all,2=A Little,3=Quite a Bit,4=Very Much). Each score range from 0 to 100 with a higher score representing a greater degree of symptoms and a worse QoL.
Time Frame: Baseline, 21 Months (EOT) up to follow-up
Population: SAS included all participants who received at least 1 administration of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 1: Imalumab 7.5 mg/kg + 5-Fluorouracil/Leucovorin (FU/LV) | Part 1: Imalumab 7.5 mg/kg + Panitumumab | Part 1: Imalumab 10 mg/kg + 5-FU/LV | Part 1: Imalumab 10 mg/kg + Panitumumab | Part 2: Imalumab 10 mg/kg + 5-FU/LV | Part 2: Standard of Care Mutant | Part 2: Imalumab 10 mg/kg + Panitumumab | Part 2: Standard of Care Wild Type
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 29 | 13 | 18 | 7
score on a scale
  Global Health Status (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 29 | 13 | 17 | 7
  Global Health Status (Baseline) | 33.33 (16.665) | 66.7 (8.335) | 75 (8.330) | 66.67 (16.665) | 68.10 (18.510) | 62.18 (25.371) | 66.18 (22.529) | 59.52 (19.501)
  Global Health Status (change from baseline (CFB)): number analyzed (Participants) | 2 | 0 | 3 | 1 | 19 | 8 | 12 | 5
  Global Health Status (change from baseline (CFB)) | 8.33 (35.355) |  | -5.56 (4.812) | -16.67 (NA) — Standard deviation was not calculated due to insufficient number of participants. | -13.16 (23.293) | -13.54 (21.333) | -10.42 (17.810) | -11.67 (9.502)
  Physical functioning scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 28 | 13 | 18 | 7
  Physical functioning scale (Baseline) | 63.33 (26.031) | 75.56 (19.249) | 88.89 (7.696) | 80 (6.670) | 78.45 (18.670) | 81.15 (15.537) | 78.89 (20.612) | 70 (17.950)
  Physical functioning scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 13 | 5
  Physical functioning scale (CFB) | 0 (0) |  | -2.22 (7.699) | -20 (NA) — Standard deviation was not calculated due to insufficient number of participants. | -5 (17.198) | -21.04 (23.489) | -4.10 (10.379) | -14.67 (15.918)
  Role functioning scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 28 | 13 | 18 | 7
  Role functioning scale (Baseline) | 50 (50) | 88.89 (19.243) | 72.22 (9.619) | 77.78 (19.243) | 74.41 (24.630) | 73.08 (30.076) | 76.85 (19.078) | 66.67 (25.459)
  Role functioning scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 13 | 5
  Role functioning scale (CFB) | -25 (35.355) |  | -16.67 (16.670) | 0 (NA) — Standard deviation was not calculated due to insufficient number of participants. | -12.04 (24.122) | -16.67 (43.642) | -11.54 (29.957) | -10 (14.910)
  Emotional functioning scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 28 | 13 | 17 | 7
  Emotional functioning scale (Baseline) | 79.67 (26.274) | 97.22 (4.809) | 91.67 (8.335) | 83.33 (16.665) | 78.87 (18.494) | 73.08 (25.720) | 77.45 (19.490) | 66.66 (18.003)
  Emotional functioning scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 12 | 5
  Emotional functioning scale (CFB) | -7 (13.675) |  | -5.56 (17.346) | -41.66 (NA) — Standard deviation was not calculated due to insufficient number of participants. | -3.24 (15.163) | -1.04 (16.925) | -2.78 (16.792) | -11.66 (20.916)
  Cognitive functioning scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 28 | 13 | 17 | 7
  Cognitive functioning scale (Baseline) | 83.33 (16.665) | 88.89 (19.243) | 100 (0) | 83.33 (16.665) | 88.10 (18.063) | 89.74 (14.496) | 93.14 (10.306) | 83.33 (23.571)
  Cognitive functioning scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 12 | 5
  Cognitive functioning scale (CFB) | 0 (0) |  | 0 (0) | -33.33 (NA) — Standard deviation was not calculated due to insufficient number of participants. | -1.85 (15.003) | -27.08 (30.779) | -8.33 (15.075) | -6.67 (9.128)
  Social functioning scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 28 | 13 | 17 | 7
  Social functioning scale (Baseline) | 77.78 (25.458) | 66.67 (0) | 77.78 (9.619) | 77.78 (9.619) | 88.69 (15.080) | 80.77 (24.387) | 73.53 (29.498) | 66.67 (27.215)
  Social functioning scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 12 | 5
  Social functioning scale (CFB) | -8.34 (11.787) |  | -22.22 (9.630) | -33.34 (NA) — Standard deviation was not calculated due to insufficient number of participants. | -13.89 (25.726) | -25 (15.430) | 0 (38.924) | -10 (19.004)
  Fatigue symptom scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 28 | 13 | 18 | 7
  Fatigue symptom scale (Baseline) | 29.67 (28.015) | 29.66 (6.351) | 22.33 (0) | 26 (6.351) | 33.74 (20.645) | 38.46 (28.580) | 29.63 (19.041) | 41.24 (21.943)
  Fatigue symptom scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 13 | 5
  Fatigue symptom scale (CFB) | 44.50 (15.797) |  | 29.45 (23.089) | 44.34 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 9.28 (19.828) | 23.63 (19.197) | 3.44 (21.919) | 13.33 (18.209)
  Nausea/vomiting symptom scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 28 | 13 | 18 | 7
  Nausea/vomiting symptom scale (Baseline) | 11.11 (19.243) | 0 (0) | 5.56 (9.624) | 16.67 (16.665) | 13.10 (22.843) | 6.41 (10.841) | 7.41 (11.746) | 4.76 (8.134)
  Nausea/vomiting symptom scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 13 | 5
  Nausea/vomiting symptom scale (CFB) | 25 (11.780) |  | 5.55 (9.619) | -16.66 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 2.78 (24.421) | 14.58 (20.773) | 5.13 (30.720) | 10 (14.906)
  Pain symptom scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 28 | 13 | 18 | 7
  Pain symptom scale (Baseline) | 38.89 (38.486) | 27.78 (9.619) | 16.67 (16.665) | 38.89 (19.243) | 31.55 (27.719) | 23.08 (30.074) | 22.22 (17.149) | 35.71 (29.546)
  Pain symptom scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 13 | 5
  Pain symptom scale (CFB) | 41.66 (35.355) |  | 11.11 (19.243) | 0 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 5.55 (21.390) | 12.50 (21.362) | 6.41 (19.882) | 13.33 (18.258)
  Dyspnea symptom scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 28 | 13 | 18 | 7
  Dyspnea symptom scale (Baseline) | 11.11 (19.243) | 11.11 (19.243) | 0 (0) | 22.22 (19.243) | 11.90 (20.716) | 20.51 (25.599) | 14.81 (26.127) | 9.52 (16.263)
  Dyspnea symptom scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 13 | 5
  Dyspnea symptom scale (CFB) | 33.34 (47.143) |  | 11.11 (19.243) | 33.33 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 5.56 (20.612) | 16.67 (30.861) | 17.95 (17.296) | 6.67 (27.886)
  Sleep disturbance/insomnia symptom scale(Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 27 | 13 | 18 | 7
  Sleep disturbance/insomnia symptom scale(Baseline) | 44.45 (38.492) | 0 (0) | 33.33 (0) | 22.22 (19.243) | 23.46 (28.964) | 20.51 (25.599) | 22.22 (25.566) | 47.62 (42.415)
  Sleep disturbance/insomnia symptom scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 17 | 8 | 13 | 5
  Sleep disturbance/insomnia symptom scale (CFB) | -0.01 (47.143) |  | 33.34 (33.335) | 0 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 7.84 (34.421) | 12.50 (30.537) | 7.69 (14.616) | -6.67 (27.886)
  Appetite loss symptom scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 28 | 13 | 18 | 7
  Appetite loss symptom scale (Baseline) | 11.11 (19.243) | 22.22 (38.492) | 11.11 (19.243) | 22.22 (19.243) | 25 (33.488) | 33.33 (38.490) | 12.96 (20.256) | 14.28 (17.816)
  Appetite loss symptom scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 13 | 5
  Appetite loss symptom scale (CFB) | 66.67 (0) |  | 33.33 (33.335) | 66.67 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 9.26 (29.826) | 4.17 (27.820) | 7.69 (24.165) | 20 (29.816)
  Constipation symptom scale (Baseline) | 11.11 (19.243) | 22.22 (19.243) | 0 (0) | 22.22 (19.243) | 17.24 (26.157) | 25.64 (30.895) | 22.22 (28.005) | 19.05 (26.227)
  Constipation symptom scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 18 | 8 | 13 | 5
  Constipation symptom scale (CFB) | 0 (0) |  | 22.22 (38.492) | 0 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 7.41 (33.442) | 16.67 (43.645) | 2.56 (34.591) | 6.67 (27.886)
  Diarrhea symptom scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 29 | 13 | 17 | 7
  Diarrhea symptom scale (Baseline) | 0 (0) | 0 (0) | 22.22 (19.243) | 11.11 (19.243) | 10.34 (18.046) | 20.51 (34.798) | 17.65 (26.660) | 23.81 (25.198)
  Diarrhea symptom scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 19 | 8 | 12 | 5
  Diarrhea symptom scale (CFB) | 33.33 (0) |  | 11.11 (19.243) | -33.33 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 8.77 (33.040) | 8.33 (38.834) | -11.11 (16.411) | 0 (23.568)
  Financial impact symptom scale (Baseline): number analyzed (Participants) | 3 | 3 | 3 | 3 | 29 | 13 | 17 | 7
  Financial impact symptom scale (Baseline) | 11.11 (19.243) | 11.11 (19.243) | 44.44 (50.918) | 44.44 (19.249) | 18.39 (30.324) | 25.64 (33.758) | 19.61 (23.743) | 28.57 (23.003)
  Financial impact symptom scale (CFB): number analyzed (Participants) | 2 | 0 | 3 | 1 | 19 | 8 | 12 | 5
  Financial impact symptom scale (CFB) | 16.67 (23.568) |  | -11.11 (19.243) | 0 (NA) — Standard deviation was not calculated due to insufficient number of participants. | -1.75 (25.996) | -12.50 (24.801) | -5.56 (12.976) | 20 (18.259)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to approximately 21 months
Description: The Medicines and Healthcare Products Regulatory Agency (MHRA) identified data integrity issues and deficiencies for AEs/SAEs for non-Shire investigational medicinal products IMPs. Per the Sponsor assessment, there was no impact of the initial non-assessment of absence of causality for SAEs associated with non-Shire IMPs (that, apart from BAX069/imalumab) on patient safety within the study, integrity of the safety conclusion or on the post-marketing safety profile for any of the non-Shire IMPs.
Arm/Group | Part 1: Imalumab 7.5 mg/kg + 5-FU/LV | Part 1: Imalumab 7.5 mg/kg + Panitumumab | Part 1: Imalumab 10 mg/kg + 5-FU/LV | Part 1: Imalumab 10 mg/kg + Panitumumab | Part 2: Imalumab 10 mg/kg + 5-FU/LV | Part 2: Standard of Care Mutant | Part 2: Imalumab 10 mg/kg + Panitumumab | Part 2: Standard of Care Wild Type
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 0/3 | 10/29 | 7/13 | 4/18 | 2/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/3 | 2/3 | 15/29 | 8/13 | 7/18 | 2/7
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 3/3 | 3/3 | 28/29 | 12/13 | 17/18 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Imalumab 7.5 mg/kg + 5-FU/LV (N=3) | Part 1: Imalumab 7.5 mg/kg + Panitumumab (N=3) | Part 1: Imalumab 10 mg/kg + 5-FU/LV (N=3) | Part 1: Imalumab 10 mg/kg + Panitumumab (N=3) | Part 2: Imalumab 10 mg/kg + 5-FU/LV (N=29) | Part 2: Standard of Care Mutant (N=13) | Part 2: Imalumab 10 mg/kg + Panitumumab (N=18) | Part 2: Standard of Care Wild Type (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 3 (3) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Imalumab 7.5 mg/kg + 5-FU/LV (N=3) | Part 1: Imalumab 7.5 mg/kg + Panitumumab (N=3) | Part 1: Imalumab 10 mg/kg + 5-FU/LV (N=3) | Part 1: Imalumab 10 mg/kg + Panitumumab (N=3) | Part 2: Imalumab 10 mg/kg + 5-FU/LV (N=29) | Part 2: Standard of Care Mutant (N=13) | Part 2: Imalumab 10 mg/kg + Panitumumab (N=18) | Part 2: Standard of Care Wild Type (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (11) | 3 (3) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 3 (3) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 4 (4) | 1 (1) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (4) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 9 (9) | 4 (4) | 3 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 5 (11) | 5 (6) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (13) | 5 (7) | 4 (9) | 1 (2)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (8) | 1 (1) | 1 (1) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 8 (9) | 2 (3) | 2 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (13) | 3 (5) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 16 (28) | 4 (11) | 5 (6) | 5 (8)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (18) | 1 (2) | 1 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venomous sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (8) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (6) | 0 (0) | 1 (1)
Blood albumin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 2 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (16) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (10) | 5 (6) | 2 (2) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (3) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 3 (4) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-Airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (22) | 2 (4)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 6 (6) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nail discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 9 (18) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trichorrhexis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
On 2016 DEC 16, the data safety monitoring board (DSMB) reviewed the periodic safety data, and in addition also reviewed available efficacy data from the first 33 PFS events and non-clinical information and recommended to terminate Study 391401.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT02448810/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT02448810/SAP_001.pdf